CLINICAL TRIAL: NCT07207772
Title: Prevention of Postoperative Pulmonary Complications in Patients Undergoing Laparoscopic Gastric Sleeve Resection by PEEP Titration Based on EIT: A Randomized Controlled Study
Brief Title: EIT-guided PEEP Titration Versus Standard Ventilation in Bariatric Surgery
Acronym: EIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jianbo Wu (Other)
Responsible Party: Sponsor-Investigator, Jianbo Wu, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YXLL-KY-2025(107)
Record Dates: First submitted 2025-09-19; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Electrical Impedance Tomography (EIT); Postoperative Pulmonary Complications (PPCs); Recruitment; Mechanical Ventilation Complication; Obesity
Keywords: Electrical Impedance Tomography (EIT); Postoperative Pulmonary Complications (PPCs); Lung protective ventilation strategy; Recruitment manoeuvre(RM); Conventional lung-protective ventilation; bariatric
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: In group P, after the titration is completed, the ventilator parameters (tidal volume, respiratory rate, and inspiratory-to-expiratory ratio) will be adjusted back to their pre-recruitment settings. Other parameters include the individualized PEEP value determined by EIT and inspiratory oxygen fraction (FiO2) of 0.5. PEEP value will be maintained throughout the surgery. The respiratory rate will be adjusted to maintain end-tidal carbon dioxide partial pressure at 35 to 45 mmHg during the operation process. A second recruitment maneuver, identical to the first, will be performed at the end of the procedure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In group C, mechanical ventilation will be administered in volume-controlled mode with a tidal volume of 8 ml/kg (based on ideal body weight). Additional settings include a PEEP of 8 cmH₂O, FiO₂ of 0.5, an inspiratory-to-expiratory ratio of 1:2, and a respiratory rate of 12 breaths/min. A recruitment maneuver (RM) will be performed 5 minutes after intubation and again after surgery, using the same protocol as in group P. The respiratory rate will be adjusted as needed to maintain end-tidal CO₂ between 35 and 45 mmHg throughout the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group P-eit (Experimental): In group P-eit, EIT electrode patches will be placed before the operation. "The Recruitment Maneuver - PEEP Titration - Recruitment Maneuver (RM-T-R) Strategy" will be implemented 5 minutes after endotracheal intubation. EIT-based optimal PEEP is defined as the crossing point of the overdistension and collapse curves during a decremental PEEP trial. Other parameters include the individualized PEEP value determined by EIT and inspiratory oxygen fraction (FiO2) of 0.5. PEEP value will be maintained throughout the surgery.All patients in the group P-eit will receive i.v. fluid loading before and a norepinephrine bolus by protocol during the RM in order to maintain a mean arterial pressure >70mm Hg and minimize the short-lasting haemodynamic depression usually observed during the RM.
  Interventions: Device: Group P-eit
- group P-8 (Active Comparator): In group P-8, mechanical ventilation will be administered in volume-controlled mode with a tidal volume of 8 ml/kg (based on ideal body weight). Additional settings include a PEEP of 8 cmH₂O, FiO₂ of 0.5, an inspiratory-to-expiratory ratio of 1:2, and a respiratory rate of 12 breaths/min. A recruitment maneuver (RM) will be performed 5 minutes after intubation and again after surgery, using the same protocol as in group P. The respiratory rate will be adjusted as needed to maintain end-tidal CO₂ between 35 and 45 mmHg throughout the procedure.
  Interventions: Device: Group P-8

INTERVENTIONS:
Device: Group P-eit — "The Recruitment Maneuver - PEEP Titration - Recruitment Maneuver (RM-T-R) Strategy" will be implemented 5 minutes after endotracheal intubation. The patient will receive an RM (peak pressure 50cm H2O, PEEP 25cmH2O, respiratory rate 6 bpm, for 10 cycles) followed by a decremental PEEP titration, during which PEEP is set to 25cm H2O and decreased stepwise by 2cm H2O every 3min until reaching 5 cmH₂O. Meanwhile, the ventilator parameters (tidal volume, respiratory rate, and inspiratory-to-expiratory ratio) will be adjusted back to their pre-recruitment settings. EIT-based optimal PEEP is defined as the crossing point of the overdistension and collapse curves during a decremental PEEP trial.
  Other Names: PEEP Titration guided by EIT
  Arms: group P-eit
Device: Group P-8 — In group p-8, mechanical ventilation will be administered in volume-controlled mode with a tidal volume of 8 ml/kg (based on ideal body weight). Additional settings include a PEEP of 8 cmH₂O, FiO₂ of 0.5, an inspiratory-to-expiratory ratio of 1:2, and a respiratory rate of 12 breaths/min. A recruitment maneuver (RM) will be performed 5 minutes after intubation and again after surgery, using the same protocol as in group P-eit. The respiratory rate will be adjusted as needed to maintain end-tidal CO₂ between 35 and 45 mmHg throughout the procedure.
  Other Names: fixed peep =8cmH2O
  Arms: group P-8

SUMMARY:
This study is a prospective, single-center, single-blind, randomized controlled clinical trial. Patients scheduled for laparoscopic bariatric surgery will be selected and randomly assigned to either the EIT-guided individualized PEEP group (Group P-eit) or the control group (Group P-8). Group P will be ventilated using the PEEP value determined by EIT, while Group C will be ventilated with a fixed PEEP value of 8 cmH2O.The primary outcome is the incidence of postoperative pulmonary complications (PPCs) within 72 hours after surgery.

DETAILED DESCRIPTION:
This is a single-center, single-blind，randomized controlled trial conducted at the First Affiliated Hospital of Shandong First Medical University in Jinan City,Shandong Province, China. This randomized controlled trial has been approved by the Ethics Committee of The First Affiliated Hospital of Shandong First Medical University (YXLL-KY-2025(107)).And it complies with the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines. A total of 118 participants will be randomly allocated to the EIT-guided individualized PEEP group (Group P ) (n = 59) or the control group (Group C) (n = 59). Recruitment for this study has begun on July 28, 2025, and will continue through the end of 2026.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years;
2. Plan to receive laparoscopic bariatric surgery under general anesthesia;
3. American Society of Anaesthesiologists (ASA) physical status I-III;
4. BMI between 30 and 55 kg/m2;
5. Voluntary participation in this study and signing of an informed consent form.

Exclusion Criteria:

1. History of smoking or previous thoracic surgery;
2. Invasive mechanical ventilation within 30 days;
3. Pregnancy;
4. Allergy to EIT electrodes;
5. Persistent hemodynamic instability or refractory shock;
6. Severe cardiopulmonary disease (e.g., severe COPD (Chronic obstructive pulmonary disease), NYHA (New York Heart Association) Class III or IV, acute coronary syndrome, or sustained ventricular tachycardia);
7. Severe pulmonary hypertension (systolic pulmonary artery pressure >40 mmHg);
8. Increased intracranial pressure, intracranial injury/tumor, or neuromuscular disorders;
9. Conversion to laparotomy;
10. Planned transfer to intensive care unit after surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative pulmonary complications | postoperative within 72 hours
  Participants who developed at least one complication are considered as meeting the primary outcome. The PPCs are defined as follows :
  1. . Pneumonia (using to the US Centres for Disease Control Criteria ;
  2. . Respiratory failure
  3. . Bronchospasm (newly detected expiratory wheezing treated with bronchodilators);
  4. . Pleural effusion
  5. . Pneumothorax
  6. . Atelectasis
  7. . Pulmonary aspiration
  8. . Cardiogenic pulmonary oedema (clinical signs of congestion, including dyspnoea, oedema, rales, and jugular venous distention, with chest X-ray demonstrating an increase in vascular markings and diffuse alveolar interstitial infiltrates).

SECONDARY OUTCOMES:
The point-of-care lung ultrasound (LUS) score | at 30 minutes after endotracheal extubation, 8:00 AM on postoperative day 1 (POD 1) and postoperative day 2 (POD2).
  The point-of-care lung ultrasound (LUS) score at 30 min after endotracheal extubation, 8:00 AM on postoperative day 1 (POD 1) and postoperative day 2 (POD2).
The severity of PPCs: | postoperative within 72 hours
  (i) None: planned use of supplemental oxygen or mechanical respiratory support as part of routine care, but not in response to a complication or deteriorating physiology. Therapies that are purely preventive or prophylactic, for example, high-flow nasal oxygen or continuous positive airway pressure (CPAP), should be recorded as none;(ii) Mild: therapeutic supplemental oxygen FiO2< 0.6. (iii) Moderate: therapeutic supplemental oxygen FiO2 ≥ 0.6, requirement for high-flow nasal oxygen, or both. (iv) Severe: unplanned non-invasive mechanical ventilation, CPAP or invasive mechanical ventilation requiring tracheal intubation.
Arterial blood gas analysis | 5 minutes post-intubation (before recruitment maneuver), 1 hour after PNP, at surgery conclusion, and 30 minutes post-extubation.
  Arterial blood gas analysis will be performed at: 5 minutes post-intubation (before recruitment maneuver), 1 hour after PNP, at surgery conclusion, and 30 minutes post-extubation.

CONTACTS AND LOCATIONS:
Overall Officials: NA GUO, MS., Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China